CLINICAL TRIAL: NCT03465917
Title: Physiological Study of the Efficacy and Mechanistic Effects of Alcohol Renal Denervation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 112014-023
Record Dates: First submitted 2018-02-20; First posted 2018-03-14 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Renal Denervation (Experimental): Renal denervation using the Peregrine Catheter for extravascular administration of ethanol
  Interventions: Combination Product: Renal Denervation

INTERVENTIONS:
Combination Product: Renal Denervation — Bilateral denervation of the renal arteries using extravascular administration of neurolytic alcohol

SUMMARY:
Hypertension is a major risk factor for heart disease and stroke, two of the leading causes of death in the United States. Hypertension is a common and widespread problem; unfortunately, current treatment strategies fail to adequately control blood pressure in up to 50% of patients either because of failure to take prescribed medications (because of cost, side effects, inconvenience etc.) or lack of therapeutic response. Indeed, it is estimated that 50% of patients stop taking antihypertensive medication within 6-12 months after the initiation of drug therapy.

Despite enthusiasm for a novel approach called renal denercation, presently there are no integrative studies of the antihypertensive effect of renal denervation on the multiple regulatory pathways it may consequentially affect. Experimental evidence from pre-clinical models suggests the effects are due to reducing efferent sympathetic activity and thus lowering blood pressure by altering the renin-angiotensin system. Uncontrolled clinical studies in humans suggest that when effective, this procedure may also lower renal sympathetic nerve activity. However the sympathetic response to monopolar radiofrequency therapy has been highly variable. Moreover, there have been no assessments of procedural efficacy performed in humans. Thus the actual mechanism by which this type of procedure reduces BP in humans is largely unknown, making it extremely difficult to identify the appropriate patients for this invasive procedure.

Recently, chemical renal denervation using ethanol (EtOH), was demonstrated to markedly lower blood pressure in small numbers of patients with resistant hypertension. However the mechanisms by which blood pressure is altered using this novel technique in humans is entirely unknown, and procedural efficacy has also not been assessed. Therefore it is unclear, whether in humans renal sympathetic nerve activity is lowered following renal denervation using this new approach. The Investigators propose to use high resolution physiological testing to determine the effects of chemical renal artery denervation on sympathetic activity.

Therefore the global objective of this physiological study is to provide the first detailed assessment of the integrated mechanistic effects of chemical renal nerve denervation in humans with hypertension that is uncontrolled by conventional treatment (because of lack of adherence or response to therapy).

DETAILED DESCRIPTION:
AIM1: The first aim of the study will be to determine the efficacy of chemical renal denervation in altering renal sympathetic nerve activity. This objective will be assessed by change in urinary catecholamines and sympathetic activity in the kidney 8 weeks post renal denervation (+/- 7 days). Specifically the investigators will compare the change in peak concentrations of 6-18F-fluorodopamine radioactivity in the renal cortex after renal denervation. A finding of a reduction in 6-18F-fluorodopamine radioactivity in the renal cortex will suggest that the chemical denervation has reduced sympathetic innervation in the kidney. The secondary assessment of efficacy will be via change in excretion of urinary norepinephrine, assessed by 24 hour urine collection. In addition, the investigators will measure plasma norepinephrine and metanephrine concentrations to isolate the systemic contribution from the kidney. Again a reduction in sympathetic innervation of the kidney by renal denervation will reduce norepinephrine excretion.

AIM 2: The second aim of the study will be to utilize high resolution physiological testing to identify how chemical renal denervation alters the integrative regulation of blood pressure. The proposal entails using classic physiological techniques to examine blood pressure regulation, which are well established in this laboratory. Briefly the testing will include a detailed assessment of hemodynamics, autonomic function, neurohormonal volume control, renal blood flow, endothelial function and vascular compliance. While mean blood pressure is the product of cardiac output × total peripheral resistance, reductions in blood pressure may be via a number of divergent mechanisms following renal denervation. Following this study, the investigators will be able to characterize how blood pressure is reduced, and whether there is individual variability in the response.

Experimental protocol. All patients will be required to undergo a battery of testing at baseline, and at 8 weeks post renal denervation. At the 8 week appointment patients will be followed up again at 6 and 12 months with an office blood pressure measurement, ambulatory blood pressure monitoring, vital signs, adverse events, assessment of renal anatomy (at 6 months and assessment of renal function.

Autonomic function testing and blood volume (Baseline, week 8): Prior to testing all patients will consume a standardized isocaloric diet provided to them for 3 days. The diet will follow the principles of the DASH diet (Dietary Approaches to Stop Hypertension). In addition, patients will avoid caffeine and alcoholic beverages for ≥24 h prior to testing, other fluid intake will be ad libitum. All studies will take place in the morning after a >12h fast. A fasting resting blood sample will be taken for measurement of FGF-23, electrolytes, hemoglobin, hematocrit, insulin and glucose. Patients will be instructed to withhold medication on the morning of this visit and a urine sample will be collected to confirm medication compliance. Autonomic function tests including spontaneous and controlled breathing, Valsalva, cold pressor test, submaximal handgrip to fatigue with post-exercise circulatory arrest, 30º and 60º head-up tilt will be performed. Measurements will include: MSNA recorded from the peroneal nerve by microneurography, beat-to-beat arterial pressure (Nexfin, BMEYE), brachial blood pressure will be measured by electrosphygmomanometry (Suntech), heart rate (HR, lead II of the ECG), cardiac output (Qc, modified acetylene rebreathing method), stroke volume (SV=Qc/HR), renal artery blood flow from doppler and total peripheral resistance (TPR=mean BP/Qc). Neurohumoral measurements include: catecholamines, plasma renin activity, aldosterone, and vasopressin will be performed at baseline and after 20 minutes of 60º head-up tilt. Sympathetic vascular transduction will be determined by the simultaneous measurement of forearm blood flow and vascular conductance (Doppler ultrasound) and MSNA at baseline. Blood volume will be measured in the sitting position by the modified carbon monoxide rebreathing technique.

Vascular, ventricular and endothelial function testing (Baseline, 8 weeks, 6 months): As systolic blood pressure is largely determined by arterial stiffness and afterload the investigators will measure the effect of renal denervation in a number of ways. Arterial stiffness will be measured using the SphygmoCor device from which the measurement of peripheral and central pulse wave velocity, augmentation index and central blood pressures will determined. In addition, based on the Windkessel model, total arterial compliance will be calculated from stroke volume/pulse pressure, effective arterial stance will be calculated from end systolic pressure/stroke volume. Aortic age, will be derived using the Modelflow method and vascular compliance as beta stiffness. Two- and three-dimensional echo for left ventricular volumes and pulse wave Doppler, Tissue Doppler parameters, and color M-Mode Doppler for assessment of diastolic function will also be performed, using a standard echo machine (Phillips, iE33). Offline analysis for torsion and strain will be performed using commercially available software (Qlab). Finally, brachial artery flow-mediated (endothelium-dependent) and nitroglycerin-induced (endothelium-independent) vasodilatation will be measured using a high-resolution Doppler ultrasound machine in the supine position.

Positron emission tomography (PET) imaging (Baseline, 8 weeks): Subjects who agree to participate in our study will travel to the National Institute of Neurological Disorders and Stroke, Bethesda Maryland, and undergo PET imaging of sympathetic activity in the kidney using PET/CT scanner (Siemens).

ELIGIBILITY:
9.1 Please indicate the inclusion criteria for enrollment: Six patients will participate in this study. Patients who present with uncontrolled hypertension (classified as clinic systolic blood pressure not at target level >140mmHg) to their primary care provider, emergency room (ER), specialist hypertension clinic or urgent care center will be asked to participate.

Inclusion criteria include:

1. Patient presents with treated or untreated hypertension.
2. Adults aged 18-75 years, male or female
3. Patient has a clinic systolic blood pressure >140mmHg (average of 3 measurements), or >135mmHg in patients with type II diabetes
4. Patient has a daytime mean systolic blood pressure of ≥135 and diastolic blood pressure ≥85mHg based on 24 hours ambulatory blood pressure monitoring
5. Investigator judges that the subject can be managed safely for up to 12 weeks (4 weeks run-in plus 8 weeks post-treatment) with the use of standard background regimen of losartan/hydrochlorothiazide; patients with true resistant hypertension will be required to maintaining current antihypertensive regime for the duration of the study.

Exclusion Criteria. Any patient who meets any of the following exclusion criteria will not be eligible for the study.

1. Patient has known or suspected secondary hypertension
2. Use of systemic drugs that may be used for the treatment of hypertension, for a non-hypertension indication for the trial, (e.g. atrial fibrillation/atrial flutter, heart failure, or calcium channel blocker for heart rate control).
3. Renal artery stenosis ≥ 50% diameter stenosis, or aneurysm(s)
4. Patients with atrial fibrillation.
5. Patient has type 1 diabetes
6. Patient has type 2 diabetes and evidence of peripheral neuropathy
7. History of previous stenting or balloon angioplasty of the renal arteries.
8. Untreated hypothyroid or hypo-parathyroid.
9. Orthostatic hypotension defined as >20 mmHg of systolic blood pressure and/or more than 10 mmHg in diastolic blood pressure fall after standing for 3mins
10. Renal artery anatomy as assessed by imaging (CT-angiogram or, MR angiogram or renal angiogram) meeting the following criteria:

    1. Single renal artery or two renal arteries, if either has a diameter of < 5 mm or > 7 mm or a length of < 11 mm,
    2. Accessory renal arteries with diameter > 2.0 mm and < 5.0 mm,
    3. Excessive renal artery tortuosity based on Investigator judgment,
    4. Moderate or severe, and diffuse renal artery calcification, and/or
    5. Renal anatomic renovascular abnormalities (as assessed by renal imaging) that would increase the risk of renal catheterization.
11. Occlusive peripheral vascular disease that would preclude percutaneous access for the procedure.
12. Patient is known to have a unilateral non-functioning kidney or unequal renal size (> 2cm difference in renal length between kidneys).
13. Single kidney, kidney tumor, urinary tract obstruction, or other anatomic abnormality. Note: Simple renal cysts are not an exclusion.
14. Previous renal denervation.
15. History of renal transplantation.
16. Estimated eGFR (by the CKD-Epi formula) ≤45 mL/min per 1.73 m2, or on chronic renal replacement therapy. Patients with eGFR of <60 mL/min per 1.73 m2 will undergo additional renal function monitoring post procedure and/or contrast exsposure.
17. Unexplained hypokalemia (i.e. K < 3.5 mEq/L in patients not on a potassium-wasting diuretic).
18. Patient in whom an ABPM device cannot be used due to arm size (>50 cm arm circumference) or other reasons as identified by the Investigator or study coordinator.
19. Patient with severe cardiac valve stenosis for which, in the opinion of the Investigator, a significant reduction of blood pressure is contraindicated.
20. Heart failure greater than asymptomatic, New York Heart Association Functional Classification, class I, stage B heart failure
21. Patient with history of myocardial infarction, unstable angina pectoris, or stroke during the 6 months prior to screening
22. Known primary or secondary pulmonary hypertension.
23. Active infection.
24. Patient requiring chronic oxygen support or has severe COPD.
25. Patient has known hypersensitivity to contrast agents that cannot be adequately pre-medicated
26. A known hypersensitivity to Dehydrated Alcohol Injection.
27. Platelet count < 75,000/microliter and/or known bleeding diathesis or coagulopathy at time of screening.
28. Receiving anticoagulant drugs (e.g., warfarin, dabigatran, rivaroxaban, apixaban, edoxaban, or low molecular weight heparins), that in the opinion of the investigator, would affect the safety of the trial procedure. Use of antiplatelet drugs such as aspirin and/or thienopyridines (e.g., clopidogrel) are permitted.
29. Patient has current problems with substance abuse (e.g. alcohol, illegal drugs, etc.).
30. Patient on high dose of steroids or immunosuppressant therapy.
31. Patient has a history of myocardial infarction, unstable angina pectoris, or stroke during the 3 months prior to screening.
32. Patients with a history of pre-eclampsia
33. patients with fibromuscular dysplasia
34. patients with history of pyelonephritis within 6 months
35. patients with history of recurrent (> one episode) kidney stones or history of kidney stones within the last year
36. Pregnant or nursing or planning to become pregnant during the trial time period.

    Note: If subject is of childbearing potential, as defined in the protocol, agrees to use of contraception.
37. Any acute or chronic condition that the investigator believes will adversely affect the ability to interpret the data or will prevent the subject from completing the trial procedures, or has a life expectancy of < 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Renal sympathetic activity | Change in renal sympathetic activity at 8 weeks
  18F-Fluorodopamine scanning of the kidney

SECONDARY OUTCOMES:
Blood pressure | Change in ambulatory blood pressure 24 hours, 1 week, 8 weeks, 6 months and 12 months after denervation.
  24-hour ambulatory blood pressure
Muscle sympathetic activity | Change in Muscle sympathetic nervous system activity 8 weeks, 6 months after renal denervation
  Muscle sympathetic nervous system activity at rest and during autonomic function testing
Vascular function | Change in flow mediated dilation 8 weeks, 6 months after renal denervation
  Flow mediated dilation
Vascular stiffness | Change in pulswave velocity at 8 weeks, 6 months after renal denervation
  Pulse wave velocity

CONTACTS AND LOCATIONS:
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hearon CMJ, Howden EJ, Fu Q, Yoo JK, Dias KA, Roberts-Reeves MA, Samels M, Sarma S, Nesbitt S, Vongpatanasin W, Goldstein DS, Addo T, Levine BD. Evidence of Reduced Efferent Renal Sympathetic Innervation After Chemical Renal Denervation in Humans. Am J Hypertens. 2021 Aug 9;34(7):744-752. doi: 10.1093/ajh/hpab022. PMID 33677553